CLINICAL TRIAL: NCT02695407
Title: Occurrence of Radial Artery Stenosis Following PICCO Catheter Cannulation
Brief Title: Radial Artery Stenosis Following PiCCO Catheter Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Magdalena Wujtewicz, assistant professor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GUMed-Wu-001
Record Dates: First submitted 2016-01-25; First posted 2016-03-01 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Artery Stenosis
Keywords: artery cannulation; haemodynamic monitoring
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 days cannulation (Experimental): radial artery cannula removed after 3 days
  Interventions: Other: 3 days cannulation
- 5 days cannulation (Experimental): radial artery cannula removed after 5 days
  Interventions: Other: 5 days cannulation

INTERVENTIONS:
Other: 3 days cannulation — assessment of artery stenosis after 3 days of artery cannulation
  Arms: 3 days cannulation
Other: 5 days cannulation — assessment of artery stenosis after 5 days of artery cannulation
  Arms: 5 days cannulation

SUMMARY:
Cardiac output monitoring devices are commonly used in ICU patients. The most precise use direct measurement, which require artery cannulation. The gold standard is Swan-Ganz catheter, but it is a very invasive technique. PiCCO (Pulse index Continuous Cardiac Output) is the alternative way of haemodynamic monitoring. This technology is the easy, less invasive and cost-efficient tool for determining the main hemodynamic parameters of critically ill patients. It is based on two physical principles - transpulmonary thermodilution and pulse contour analysis. Both principles allow the calculation of haemodynamic parameters in critically ill patients. PiCCO method requires peripheral artery cannulation.

Cannulation may be followed by artery stenosis.

Aims of the study are:

1. to verify the occurrence of radial artery stenosis after 3 days of having a PiCCO cannula in place.
2. whether 5 days cannulation of radial artery with PiCCO catheter is related to more frequent stenosis rate.

An additional assessment:

1. to check whether the eventual stenosis is still present after 3, 14 and 30 days after decannulation - assessment depending on patients availability

DETAILED DESCRIPTION:
Barbeau test and Doppler - ultrasonography preceded radial artery cannulation. Catheter removal (after 3 or 5 days of cannulation) is followed by Doppler - usg. Usg -Doppler is performed also 3, 14 and 30 days after decannulation - depending on patient being available

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients with haemodynamic monitoring required

Exclusion Criteria:

* Barbeau test type D in radial artery
* artery inaccessible for cannulation - based on doppler ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with artery stenosis after radial artery decannulation, confirmed by Doppler ultrasonography | up to 5 days after cannulation
  in one group usg, following decannulation will be performed 3 days after cannulation, in the second group - decannulation and usg will be done 5 days after cannulation.

SECONDARY OUTCOMES:
Number of patients with persistent artery stenosis after radial artery decannulation, confirmed by Doppler ultrasonography | 3, 14 and 30 days after decannulation
  usg will be performed 3, 14 and 30 days after decannulation; depending on patients availability

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Wujtewicz, Principal Investigator — Department of Ophthalmology, Mediacal University of Gdansk, Gdansk, Poland
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

REFERENCES:
- [Derived] Wujtewicz M, Regent B, Marszalek-Ratnicka R, Smugala A, Szurowska E, Owczuk R. The Incidence of Radial Artery Occlusion in Critically Ill Patients after Cannulation with a Long Catheter. J Clin Med. 2021 Jul 19;10(14):3172. doi: 10.3390/jcm10143172. PMID 34300338